CLINICAL TRIAL: NCT02787187
Title: A Prospective Randomized Controlled Study Comparing Standard and Extended Lymphadenectomy for Pancreatic Head Cancer
Brief Title: Lymphadenectomy for Pancreatic Head Cancer: Standard or Extended?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Weishen WANG, Doctor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBP-RCT-001
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Standard lymphadenectomy; extended lymphadenectomy; pancreaticoduodenectomy
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard resection (Active Comparator): Pancreaticoduodenectomy (child's digestive reconstruction); Standard lymphadenectomy: No 5 6 8a 12b1 12b2 12c 13a 13b 14a 14b 17a 17b
  Interventions: Procedure: Pancreaticoduodenectomy with Standard lymphadenectomy
- Extended resection (Experimental): Pancreaticoduodenectomy (child's digestive reconstruction)extended lymphadenectomy No8p 12a 12p 14c 14d 16
  Interventions: Procedure: Pancreaticoduodenectomy with Extended lymphadenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy with Standard lymphadenectomy — Pancreaticoduodenectomy：child's digestive reconstruction standard lymphadenectomy: No 5 6 8a 12b1 12b2 12c 13a 13b 14a 14b 17a 17b
  Arms: Standard resection
Procedure: Pancreaticoduodenectomy with Extended lymphadenectomy — Pancreaticoduodenectomy：child's digestive reconstruction extended lymphadenectomy: No8p 12a 12p 14c 14d 16
  Arms: Extended resection

SUMMARY:
The purpose of this study is to compare outcomes of patients undergoing standard or extended lymphadenectomy in pancreaticoduodenectomy for pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of pancreatic ductal adenocarcinoma
* Signed the informed consents

Exclusion Criteria:

* Pathologic diagnosis of other pancreatic cancers
* Pre-operative anti-cancer treatment
* Recurrence patients
* Patients with contraindication(hepatic/ respiratory/ renal dysfunction, etc )
* Pre operative exam: Total bilirubin more than 250µmol/L
* AJCC stage IV
* Operation non radical

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 3yrs post-operation

SECONDARY OUTCOMES:
all-cause mortality | 1yr post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong SHEN, Study Director — Shanghai Ruijin Pancreatic Disease Center
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided